CLINICAL TRIAL: NCT06821139
Title: Impact of COVID-19 Pandemic on Patterns and Predictors of Intraoperative Lung Protective Ventilation in a Large Canadian Health Authority.
Brief Title: Impact of COVID-19 Pandemic on Intraoperative Ventilation Practices in Western Canada
Status: Completed | Type: Observational
Sponsor: Perseus Missirlis (Other)
Collaborators: University of British Columbia (Other)
Responsible Party: Sponsor-Investigator, Perseus Missirlis, Clinical instructor, staff anesthesiologist, Fraser Health
Organization: Fraser Health (Other)
Other Study IDs: FHREB 2020-083; H20-01683 (Other: University of British Columbia)
Record Dates: First submitted 2025-01-14; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Lung Protective Ventilation; Intraoperative Ventilation; COVID; COVID - 19; Non-cardiac Surgery
Keywords: lung protective ventilation; intraoperative ventilation; Canadian; COVID; non-cardiac surgery; predictors
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-COVID cohort: Before January 2020. The investigators considered before January 2020 as the pre-COVID era, and after June 2020 as the COVID era. The former cutoff was chosen as January 2020 contained the first COVID case in British Columbia, the province containing the study sites. The latter cutoff was chosen as it constitutes three months after March 2020, when the World Health Organization (WHO) announced COVID's pandemic status, and British Columbia announced a state of emergency with the start of isolation policies. The investigators hypothesized that any impact of the COVID pandemic on lung protective ventilation practice patterns would unlikely to have occurred prior COVID's arrival in BC, but would likely be in full swing three months after initiation of widespread social isolation, a very palpable event in society.
- New normal cohort: After June 2020. The investigators considered before January 2020 as the pre-COVID era, and after June 2020 as the COVID era. The former cutoff was chosen as January 2020 contained the first COVID case in British Columbia, the province containing the study sites. The latter cutoff was chosen as it constitutes three months after March 2020, when the WHO announced COVID's pandemic status, and British Columbia announced a state of emergency with the start of isolation policies. The investigators hypothesized that any impact of the COVID pandemic on lung protective ventilation practice patterns would unlikely to have occurred prior COVID's arrival in BC, but would likely be in full swing three months after initiation of widespread social isolation, a very palpable event in society.

SUMMARY:
The goal of this observational study is to ascertain the practice patterns and predictors in performing lung protective ventilation as per clinical guidelines for adult patients undergoing non-cardiac surgery in Fraser Health Authority, a large Canadian authority in the lower mainland of British Columbia, Canada. In particular, the investigators explore changes before/after the COVID-19 pandemic. The main questions it aims to answer are:

* In this population, what is the general compliance rate to lung protective ventilation
* In this population, what are the predictors of compliance before/after the COVID-19 pandemic.

This is a retrospective study using linked patient data from two databases in the health region: the anesthesia informational management system for intraoperative data, and the electronic medical record for perioperative data.

Rationale for study:

Breathing problems after surgery affect 5% to 33% of patients and can lead to serious issues like lung infections, breathing failure, and longer hospital stays, with up to a 20% risk of death within 30 days for serious cases. A proven way to reduce these risks is lung protective ventilation (LPV), a technique used during surgery where the ventilator delivers smaller breaths based on clinical guidelines and calculated using a person's ideal body weight, while applying gentle pressure to keep the lungs slightly open. While this approach has been widely adopted in intensive care units over the past 20 years, it's less commonly used in operating rooms, with fewer than half of surgeries using it. Barriers include suboptimal default ventilator settings, patients at extremes of weight, and misunderstandings of LPV among clinicians. During the COVID-19 pandemic, LPV use increased for patients with COVID-related lung problems, showing improved survival rates in ICUs. However, it's unclear if this practice carried over to surgical patients at-large or continued after the pandemic. Most studies on LPV during surgery have been conducted outside Canada, where healthcare practices and education may differ from within Canada. To address these gaps, the investigators aim to study LPV use during surgery in a large Canadian health system, identify factors that influence its use, and examine trends during and after the COVID pandemic. This research will help improve patient care by promoting the use of this effective technique in Canadian operating rooms.

DETAILED DESCRIPTION:
This observational study aims to elucidate the patterns and predictors of intraoperative lung protective ventilation (LPV) in adult patients undergoing non-cardiac surgery at Fraser Health Authority, a large Canadian health authority on the west coast of Canada, between 2014-2023. It also assesses the impact of pre-COVID vs. new-normal era on LPV compliance, and interactions of predictors with pre-COVID vs. new-normal era. LPV is defined as both 1) tidal volume of 6-8mL/kg ideal body weight and 2) positive end-expiratory pressure of 5 cmH2O or more. Intraoperative data will be derived from the intraoperative anesthesia information management system, and the perioperative data from the regional electronic medical record. The investigators will use a predictive logistic regression model to ascertain statistically significant predictors to LPV. Hypothesized predictors of LPV compliance based on literature and expert opinion will be considered for inclusion in the model. Pre-COVID and "new normal" data will be compared, and interactions with predictors will be explored. As a secondary analysis, a Shewhart chart will be used to elucidate any special cause variation in LPV compliance introduced by the COVID pandemic. For details of descriptive analyses, model derivation, and Shewhart chart methodology, please refer to study protocol.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 18
* underwent general anesthesia with endotracheal tube placement for a procedure lasting ≥30 minutes.
* included in both our clinical anesthesia record database and the National Surgical Quality Improvement Program (NSQIP) database, and linkable by usual identifiers (name, date of birth, medical record number, personal health number, date of surgery)

Exclusion Criteria:

* no endotracheal tube utilized
* cardiothoracic surgery
* organ donation surgery
* organ transplant recipient
* Hyperthermic intraperitoneal chemotherapy
* surgical procedure related to an occurrence or complication of prior procedure during the same admission/within 30 days,
* multiple NSQIP assessed cases within 30 days only for same patient
* cases in clinical anesthesia record database that are unable to be linked to NSQIP data or vice versa.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from January 2014 to December 2023, age above 18, undergoing non-cardiac and non-thoracic surgery for greater than 30 minutes with an endotracheal tube placed. Both inpatients and outpatients are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 28700 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Lung protective ventilation compliance | For patients not ventilated preoperatively: from insertion to removal of endotracheal tube (or until end of case if tube not removed). For already ventilated patients: from start to end of operation.
  Compliance with ventilation guidelines is defined as meeting two criteria. The first is that their average tidal volume is 6-8 mL/kg ideal body weight and the second is that the average positive end expiratory pressure is at least 5 cm H2O. Patients ventilated according to one or neither of the above criteria will not be considered to have been ventilated according to established guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Perseus Missirlis, MD, MSc, Principal Investigator — University of British Columbia
Locations (1):
- Fraser Health Authority, Surrey, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
Individual patient data (IPD) is obtained from medical record registries at Fraser Health Authority. While IPD used in this study will not be shared, these data (and similar data at other time frames) are freely available to investigators of subsequent proposed studies, in collaboration with an investigator at Fraser Health Authority, through the usual data access application mandated by Fraser Health Authority.

REFERENCES:
- [Background] Bender SP, Paganelli WC, Gerety LP, Tharp WG, Shanks AM, Housey M, Blank RS, Colquhoun DA, Fernandez-Bustamante A, Jameson LC, Kheterpal S. Intraoperative Lung-Protective Ventilation Trends and Practice Patterns: A Report from the Multicenter Perioperative Outcomes Group. Anesth Analg. 2015 Nov;121(5):1231-9. doi: 10.1213/ANE.0000000000000940. PMID 26332856
- [Background] Parks DA, Short RT, McArdle PJ, Liwo A, Hagood JM, Crump SJ, Bryant AS, Vetter TR, Morgan CJ, Beasley TM, Jones KA. Improving Adherence to Intraoperative Lung-Protective Ventilation Strategies Using Near Real-Time Feedback and Individualized Electronic Reporting. Anesth Analg. 2021 May 1;132(5):1438-1449. doi: 10.1213/ANE.0000000000005481. PMID 33724961
- [Background] Blum JM, Maile M, Park PK, Morris M, Jewell E, Dechert R, Rosenberg AL. A description of intraoperative ventilator management in patients with acute lung injury and the use of lung protective ventilation strategies. Anesthesiology. 2011 Jul;115(1):75-82. doi: 10.1097/ALN.0b013e31821a8d63. PMID 21552117
- [Background] Kim SH, Na S, Lee WK, Choi H, Kim J. Application of intraoperative lung-protective ventilation varies in accordance with the knowledge of anaesthesiologists: a single-Centre questionnaire study and a retrospective observational study. BMC Anesthesiol. 2018 Apr 2;18(1):33. doi: 10.1186/s12871-018-0495-7. PMID 29606090
- [Background] Young CC, Harris EM, Vacchiano C, Bodnar S, Bukowy B, Elliott RRD, Migliarese J, Ragains C, Trethewey B, Woodward A, Gama de Abreu M, Girard M, Futier E, Mulier JP, Pelosi P, Sprung J. Lung-protective ventilation for the surgical patient: international expert panel-based consensus recommendations. Br J Anaesth. 2019 Dec;123(6):898-913. doi: 10.1016/j.bja.2019.08.017. Epub 2019 Oct 3. PMID 31587835
- [Background] Guay J, Ochroch EA, Kopp S. Intraoperative use of low volume ventilation to decrease postoperative mortality, mechanical ventilation, lengths of stay and lung injury in adults without acute lung injury. Cochrane Database Syst Rev. 2018 Jul 9;7(7):CD011151. doi: 10.1002/14651858.CD011151.pub3. PMID 29985541
- [Background] Canet J, Gallart L, Gomar C, Paluzie G, Valles J, Castillo J, Sabate S, Mazo V, Briones Z, Sanchis J; ARISCAT Group. Prediction of postoperative pulmonary complications in a population-based surgical cohort. Anesthesiology. 2010 Dec;113(6):1338-50. doi: 10.1097/ALN.0b013e3181fc6e0a. PMID 21045639

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-24): https://cdn.clinicaltrials.gov/large-docs/39/NCT06821139/Prot_SAP_000.pdf